CLINICAL TRIAL: NCT06272656
Title: Evaluation of AKR1B10 as a New Marker for Interventional Therapy of Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Principal Investigator, Yuemin Nan, Director of Hepatology Department of integrated Chinese and Western Medicine, Hebei Medical University Third Hospital
Other Study IDs: AKR-TACE-001
Record Dates: First submitted 2024-01-18; First posted 2024-02-22 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: AKR1B10
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples from liver cancer patients at 4 ℃, 4000g, centrifuge for 10 minutes, and take 500 samples μ Place L in a 1.5mL EP tube and freeze at -80 ℃ for later use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC Patients treated with TACE: HCC patients who have received initial diagnosis and treatment in our hospital and are planning to receive TACE.

SUMMARY:
Primary liver cancer is currently the fourth most common malignant tumor and the second leading cause of tumor mortality in China, posing a serious threat to the lives and health of the Chinese people . At present, non-surgical treatment methods are often used, such as radiofrequency ablation (RFA), Transcatheter arterial chemoembolization (TACE), radiation therapy, and systemic anti-tumor therapy. However, whether it is surgical treatment or non-surgical treatment, commonly used liver cancer related biomarkers in clinical practice during the evaluation of treatment efficacy or regular follow-up of patients include AFP, AFP-L3%, DCP, etc. , but there are no reports on whether AKR1B10 can be used for the efficacy evaluation of these treatment methods.Therefore, this project aims to explore the clinical value of AKR1B10 in evaluating the efficacy of liver cancer treatment.

DETAILED DESCRIPTION:
Patients with hepatocellular carcinoma (HCC) treated with transarterial chemoembolisation (TACE) are enrolled in this clinical trial. In the early stage, a research team detected the levels of AKR1B10 in serum samples from 477 normal individuals, 107 benign liver tumors, 32 patients with chronic hepatitis B, 78 patients with liver cirrhosis, and 482 patients with liver cancer, and evaluated its early diagnostic value in liver cancer. It was found that AKR1B10 protein, as a serum marker for liver cancer, had significantly better performance than AFP, mainly reflected in three aspects: first, it is more sensitive, The normal background level (reference range) of AKR1B10 is significantly lower than AFP, which means that during clinical testing, changes in serum concentration are more pronounced, making it easier to identify asymptomatic early liver cancer patients; Secondly, it is more specific and has a higher detection rate for liver cancer, with lower false positive and false negative rates. In addition, more than 70% of liver cancer patients who test negative for AFP will be tested positive for AKR1B10, resulting in lower rates of missed diagnosis and misdiagnosis; Thirdly, the time to reflect changes in the condition is 6-7 times faster than AFP. The half-life of AKR1B10 is 23 hours, while AFP has a half-life of 6-7 days.This project mainly aims to explore the clinical value of AKR1B10 in evaluating the efficacy of liver cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80
* diagnosis of HCC according the AASLD criteria
* TACE is planned
* resection is impossible
* No significant underlying medical illness affecting patient's survival
* Patients available for regular follow-up according to the study protocol

Exclusion Criteria:

* Previous history of other tumors;
* Combined with other tumors;
* Received external treatment before admission;
* Patients who have received blood transfusions within one month;
* The patient was unable to participate in this study for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants have signed an informed consent form, agreeing that their samples and related information can be used for all medical studies.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
comparison of liver cancer markers AKR1B10, AFP, AFP-L3% and DCP before and after TACE | baseline, 1 month and 3 months
  Liver cancer markers AKR1B10, AFP, AFP-L3 and DCP are measured before TACE, 1 month and 3 months after TACE in order to evaluate the course of these markers after the intervention

SECONDARY OUTCOMES:
long-term survival (1-year, 3-year, 5-year) | up to 5 years
  Patients with low AKR1B10 levels have a higher survival rate
progression- free - time | up to 5 years
  Patients with low AKR1B10 levels have a longer progression- free - time

CONTACTS AND LOCATIONS:
Overall Officials: Yuemin Nan, Principal Investigator — Hebei Medical University Third Hospital
Locations (1):
- HebeiMUTH, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Zhu XD, Huang C, Shen YH, Ji Y, Ge NL, Qu XD, Chen L, Shi WK, Li ML, Zhu JJ, Tan CJ, Tang ZY, Zhou J, Fan J, Sun HC. Downstaging and Resection of Initially Unresectable Hepatocellular Carcinoma with Tyrosine Kinase Inhibitor and Anti-PD-1 Antibody Combinations. Liver Cancer. 2021 Jul;10(4):320-329. doi: 10.1159/000514313. Epub 2021 Mar 30. PMID 34414120
- [Background] Wang Z, Ren Z, Chen Y, Hu J, Yang G, Yu L, Yang X, Huang A, Zhang X, Zhou S, Sun H, Wang Y, Ge N, Xu X, Tang Z, Lau W, Fan J, Wang J, Zhou J. Adjuvant Transarterial Chemoembolization for HBV-Related Hepatocellular Carcinoma After Resection: A Randomized Controlled Study. Clin Cancer Res. 2018 May 1;24(9):2074-2081. doi: 10.1158/1078-0432.CCR-17-2899. Epub 2018 Feb 2. PMID 29420221
- [Result] Tateishi R, Shiina S, Yoshida H, Teratani T, Obi S, Yamashiki N, Yoshida H, Akamatsu M, Kawabe T, Omata M. Prediction of recurrence of hepatocellular carcinoma after curative ablation using three tumor markers. Hepatology. 2006 Dec;44(6):1518-27. doi: 10.1002/hep.21408. PMID 17133456
- [Result] Yoo J, Lee MW, Lee DH, Lee JH, Han JK. Evaluation of a serum tumour marker-based recurrence prediction model after radiofrequency ablation for hepatocellular carcinoma. Liver Int. 2020 May;40(5):1189-1200. doi: 10.1111/liv.14406. Epub 2020 Mar 13. PMID 32056353
- [Result] Ye X, Li C, Zu X, Lin M, Liu Q, Liu J, Xu G, Chen Z, Xu Y, Liu L, Luo D, Cao Z, Shi G, Feng Z, Deng H, Liao Q, Cai C, Liao DF, Wang J, Jin J, Cao D. A Large-Scale Multicenter Study Validates Aldo-Keto Reductase Family 1 Member B10 as a Prevalent Serum Marker for Detection of Hepatocellular Carcinoma. Hepatology. 2019 Jun;69(6):2489-2501. doi: 10.1002/hep.30519. Epub 2019 Apr 6. PMID 30672601
- See also: Pubmed — https://pubmed.ncbi.nlm.nih.gov

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-12-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT06272656/Prot_ICF_000.pdf